CLINICAL TRIAL: NCT06623526
Title: An Open-label, Randomized, Fasting, Single-Crossover Study to Compare the Pharmacokinetic Interactions and Safety of YHR2402 Monotherapy and YHR2402 and YHR2403 Co-Administration in Healthy Volunteers
Brief Title: Clinical Trial to Evaluate the PK Interactions of YHR2402 Monotherapy and YHR2402 and YHR2403 Co-Administration in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yuhan Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: YHP2401-101
Record Dates: First submitted 2024-09-30; First posted 2024-10-02 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Healthy Volunteers
Keywords: pharmacokinetic interactions; Drug-Drug Interaction

STUDY DESIGN:
Intervention Model Description: two-way crossover
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sequence Group 1 (Experimental): 13 subjects, Cross-over, Single dose of YHR2402 on day 1, Co-Administration of YHR2402 and YHR2403 on day 15
  Interventions: Drug: YHR2402; Drug: YHR2402+YHR2403
- Sequence Group 2 (Experimental): 13 subjects, Cross-over, Co-Administration of YHR2402 and YHR2403 on day 1, Single dose of YHR2402 on day 15
  Interventions: Drug: YHR2402; Drug: YHR2402+YHR2403

INTERVENTIONS:
Drug: YHR2402 — Test Drug: YHR2402
Drug: YHR2402+YHR2403 — Test Drug: YHR2402+YHR2403

SUMMARY:
An open-label, randomized, single-dose, crossover study to evaluate the pharmacokinetic interactions and safety after co-administration of YHR2402 and YHR2403 compared to the administration of YHR2402 independently in healthy subjects

DETAILED DESCRIPTION:
26 healthy subjects will be randomized to one of the 2 groups in the same ratio.

"YHR2402" and "YHR2402"+"YHR2403" will be administered to Subjects in group 1 by crossover design on day 1, 15

"YHR2402"+"YHR2403" and "YHR2402" will be administered to Subjects in group 2 by crossover design on day 1, 15.

ELIGIBILITY:
Inclusion Criteria:

* Those who are 19 years old and under 55 years old at the screening visit
* Those whose weight is over 50kg(male), over 45kg(female) and their body mass index (BMI) shall be between 18.0 kg/m2 and 30.0 kg/m2
* Those who express their voluntary consent to participate in the trial by signing a written consent
* Those who are judged eligible to participate in the trial by the principal investigator(or delegated investigators) after screening test

Exclusion Criteria:

* Those who have participated in a bioequivalence study or other clinical trials and have been administered with investigational products in 6 months prior to the first administration
* Others who are judged ineligible to participate in the trial by the principal investigator

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2024-10-04 (Actual); Primary Completion 2024-11-06 (Actual); Study Completion 2024-11-11 (Actual)

PRIMARY OUTCOMES:
Area under the plasma drug concentration-time curve [AUCt] | 0-96 hours
  of Chlorpheniramine, Dihydrocodeine and Dl-Methylephedrine
Maximum plasma concentration [Cmax] | 0-96 hours
  of Chlorpheniramine, Dihydrocodeine and Dl-Methylephedrine

SECONDARY OUTCOMES:
Area under the plasma drug concentration-time curve from time 0 to infinity [AUCinf] | 0-96 hours
  of Chlorpheniramine, Dihydrocodeine and Dl-Methylephedrine
Area under the plasma drug concentration-time curve/Area under the plasma drug concentration-time curve from time 0 to infinity [AUCt/AUCinf] | 0-96 hours
  of Chlorpheniramine, Dihydrocodeine and Dl-Methylephedrine
Time of Maximum observed plasma concentration [Tmax] | 0-96 hours
  of Chlorpheniramine, Dihydrocodeine and Dl-Methylephedrine
Apparent Terminal Elimination Half-life [t1/2] | 0-96 hours
  of Chlorpheniramine, Dihydrocodeine and Dl-Methylephedrine

CONTACTS AND LOCATIONS:
Overall Officials: Mingul Kim, Principal Investigator — Jeonbuk National University Hospital
Locations (1):
- Jeonbuk National University Hospital, Jeonju, South Korea

IPD SHARING:
Plan to Share IPD: No